CLINICAL TRIAL: NCT00021424
Title: Phase I/Pilot Study of Intralesional Immunotherapy With A Recombinant Avipox Virus Engineered To Express A Triad Of Co-Stimulatory Molecules In Patients With Advanced Squamous Cell Carcinoma Of The Head And Neck
Brief Title: Vaccine Therapy in Treating Patients With Stage IV Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068782; NCI-01-DC-0006; NCI-3210; NCT00006410 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2002-08

CONDITIONS: Head and Neck Cancer; Metastatic Cancer
Keywords: stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; skin metastases
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasm Metastasis; Squamous Cell Carcinoma of Head and Neck

INTERVENTIONS:
Biological: recombinant fowlpox-TRICOM vaccine

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy in treating patients who have stage IV head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and dose-limiting toxic effects of recombinant fowlpox-TRICOM vaccine in patients with advanced squamous cell carcinoma of the oral cavity or oropharynx or nodal or dermal metastases.
* Determine the safety profile of this regimen in these patients.
* Determine the clinical activity of this regimen, in terms of inflammation at injection site(s) and disease regression or stabilization, in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive recombinant fowlpox-TRICOM vaccine (rF-TRI) intralesionally once on weeks 0, 3, and 8. Beginning on week 16, patients may receive additional rF-TRI once every 8 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of rF-TRI until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 1 year.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV squamous cell carcinoma of the oral cavity or oropharynx or nodal or dermal metastases for which current available treatment is not likely to offer a survival advantage or result in significant palliation

  * Unresectable locoregional recurrence after maximum radiotherapy OR
  * Local disease with unresectable distant metastases involving:

    * Base of skull
    * Prevertebral fascia
    * Deep neck muscles
    * Carotid artery (requiring resection)
    * Nasopharynx and/or pterygoid muscles
* Ineligible to receive radiotherapy to head and neck during study
* Primary intraoral lesions must be measurable and accessible to intralesional injections
* No metastatic brain lesions, cerebral metastasis, or leptomeningeal disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-2

Life expectancy:

* At least 2 months

Hematopoietic:

* Absolute neutrophil count greater than 1,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 8 g/dL

Hepatic:

* Bilirubin less than 1.5 mg/dL
* AST/ALT less than 4 times upper limit of normal (ULN)
* PT/PTT less than 1.5 times ULN

Renal:

* Creatinine less than 2.0 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No evidence of congestive heart failure
* No serious cardiac dysrhythmia
* No evidence of recent prior myocardial infarction on EKG
* No clinical coronary artery disease

Neurologic:

* No history of seizures or concurrent seizure disorder
* No evidence of encephalitis, multiple sclerosis, or other structural brain lesion(s) by clinical or radiological evaluation

Immunologic:

* No risk of immune system compromise
* HIV negative
* No hypersensitivity to eggs
* No significant history of allergies (e.g., anaphylaxis or angioedema)

Other:

* No active or chronic infection
* No other serious concurrent medical illness
* No other malignancy unless previously treated with curative intent and no evidence of persistent or recurrent disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered

Chemotherapy:

* No more than 2 prior chemotherapy regimens
* At least 4 weeks since prior chemotherapy and recovered

Endocrine therapy:

* At least 4 weeks since prior systemic corticosteroids
* No concurrent systemic corticosteroids

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy to more than 50% of nodal groups

Surgery:

* More than 4 weeks since prior surgery for primary or metastatic lesions and recovered
* No prior splenectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-06

CONTACTS AND LOCATIONS:
Overall Officials: Susan Rudy, MSN, Study Chair — National Institute on Deafness and Other Communication Disorders (NIDCD)
Locations (1):
- Warren Grant Magnuson Clinical Center, Bethesda, Maryland, United States